CLINICAL TRIAL: NCT03474731
Title: Clinic to Community Navigation to Improve Diabetes Outcomes
Acronym: CCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nancy Schoenberg (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Nancy Schoenberg, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0314-P6H; R01DK112136 (NIH)
Record Dates: First submitted 2017-10-11; First posted 2018-03-23 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Background and justification: Nearly 29 million Americans (9.3% of the population) have type 2 Diabetes Mellitus (T2DM) and another 86 million are considered prediabetic, 20-30% of whom will develop diabetes within five years.4,5 T2DM disproportionately affects those from lower socioeconomic status (SES) and rural backgrounds. Appalachian residents represent an extreme version of this already vulnerable population, with rates of diabetes 46% higher than national averages.6,7 We have developed, pilot tested (N=41) and refined (N=48 in-depth interviews, 4 focus groups with 31 participants, and 2 CAB meetings with 16 members), a culturally appropriate, feasible, and promising intervention that combines diabetes self-management education and tailored patient navigation intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diabetes Self-Management Program (DSMP) only (Experimental): group education classes of the Diabetes Self-Management Program, (DSMP)
  Interventions: Behavioral: Diabetes Self-Management Program (DSMP)
- Tailored Patient Navigation (PN) only (Experimental): assisting patients in navigation to physician offices, allowing for standard of care to follow.
  Interventions: Behavioral: Tailored Patient Navigation (PN) only
- DSMP AND Tailored Patient Navigation (Experimental): Both group education classes and patient navigation
  Interventions: Behavioral: DSMP AND Tailored Patient Navigation
- Diabetes Self-Management Program (DSMP) Delayed (Active Comparator): group education classes of the Diabetes Self-Management Program, (DSMP)
  Interventions: Behavioral: Diabetes Self-Management Program (DSMP) Delayed

INTERVENTIONS:
Behavioral: Diabetes Self-Management Program (DSMP) — The the Diabetes Self Management Program (DSMP) in a group setting: participants will attend a six week, evidence-based diabetes home self-management program. The goal of this arm of the project is to try to get participants to engage in better diabetes self-care (blood glucose testing, medication taking, diet, exercise, stress reduction, etc.).
  Participants will complete biometric data and surveys at 3, 6, and 9 months post randomization.
  Arms: Diabetes Self-Management Program (DSMP) only
Behavioral: Tailored Patient Navigation (PN) only — Tailored Patient Navigation (PN) only: trained Community Health Workers (CHW) will meet one-on-one with participants to assess the barriers experienced in adhering to medical appointments and will implement a navigation program accordingly.
  The goal of this arm of the project is to try to get participants to attend recommended medical appointments. PN has been shown to improve health behavior and increase self-efficacy, all with low costs.
  Arms: Tailored Patient Navigation (PN) only
Behavioral: DSMP AND Tailored Patient Navigation — DSMP AND Tailored Patient Navigation : patient navigation followed by 6 weeks of DSMP classes after the 3 month post-test interview.
  Other Names: Clinic to Community Navigation (CCN)
  Arms: DSMP AND Tailored Patient Navigation
Behavioral: Diabetes Self-Management Program (DSMP) Delayed — Groups randomized to DSMP Delayed will receive 6 weeks of DSMP classes after the 3 month post-test interview.
  Participants will complete biometric data and surveys at 3, 6, and 9 months post randomization.
  Arms: Diabetes Self-Management Program (DSMP) Delayed

SUMMARY:
Background and justification: Nearly 29 million Americans (9.3% of the population) have type 2 Diabetes Mellitus (T2DM) and another 86 million are considered prediabetic, 20-30% of whom will develop diabetes within five years.4,5 T2DM disproportionately affects those from lower socioeconomic status (SES) and rural backgrounds. Appalachian residents represent an extreme version of this already vulnerable population, with rates of diabetes 46% higher than national averages.6,7 The investigators have developed, pilot tested (N=41) and refined (N=48 in-depth interviews, 4 focus groups with 31 participants, and 2 CAB meetings with 16 members), a culturally appropriate, feasible, and promising intervention that combines diabetes self-management education and tailored patient navigation intervention., Goal: Our goal focuses on reducing HbA1c, BMI, blood pressure, lipids, and waist circumference and improving T2DM self-management and clinic attendance. Leveraging local assets, including faith communities, local health facilities, trained community health workers, and social support, the investigators will expand a promising and refined pilot study and assess outcomes, satisfaction and cost effectiveness. Innovation and impact: The proposed project is among the first RCT to combine the two most influential approaches to diabetes control-- self-management education and tailored patient navigation in a community setting. The Community to Clinic Navigation (CCN) intervention has the potential to sustainably empower hard to reach populations with effective self-management education and enhance the quality of healthcare in traditionally underserved communities, greatly improving T2DM outcomes.

DETAILED DESCRIPTION:
1. Background: Appalachian residents maintain disproportionately high rates of Type 2 Diabetes Mellitus (T2DM) and suffer tremendous burdens from diabetic complications. The main challenges to stemming adverse outcomes from T2DM involve ensuring optimal clinical care and self-management. Because the prevalence of diabetes has tripled since 2005, the already low supply of primary care physicians combined with this tremendous chronic disease burden places huge demands on providers in rural Appalachia. Enhancing the quality and efficiency of these practices by linking to community health workers has the potential of mitigating the adverse effects of these shortages.

   Patient navigation, particularly a clinic to community navigation (CCN) model offers an innovative approach to address these inequities. Patient navigation has been implemented almost exclusively in the cancer setting, despite being promising for chronic disease management. The proposed project is, to our knowledge, the first to test a hybrid model of clinic (health promotion professional) plus community (community health worker) navigation among rural residents. Clinical patient navigation has been shown to facilitate appointment setting and return visits, may improve goal setting, and enhances some adherence (medication taking, blood glucose testing), but does not address some key psychosocial (self-efficacy, patient activation) and practical concerns (transportation, childcare, self-management) challenges. Community-based navigation programs have been shown to enhance self-efficacy, decrease community barriers to care (e.g., transportation), and improved self-management, but may be less effective in ensuring return visits and working collaboratively with the doctor.
2. Objectives: The investigators aim to test a CCN program that may improve the most salient influences on diabetes outcomes and self-management, the health care context and the patient's home context. Specifically, the investigators will (1) recruit 1200 participants from community settings with T2DM and HbA1c levels between 9-11% and randomize them to one of three arms, DSMP; PN, or combined CCN intervention; (2) the investigators will administer three quantitative assessments. All activities will take place in Appalachia. Outcomes include physiologic data (HbA1C levels, blood pressure, lipids, waist circumference and BMI, obtained by research staff); quantitative data collection of self-management (medication taking, blood glucose, appointment adherence, diet, physical activity, foot and eye care, obtained by interviewer); and psychosocial variables (self-efficacy, patient activation, obtained by interviewer).
3. Study Design: Behavioral randomized controlled trial, single blind design.
4. Study Population: Eligibility criteria: Adults 18+; Appalachian residence, and HBA1c levels between 9-11%. Those who do not meet these inclusion criteria, are cognitively impaired, or who do not wish to participate will be excluded. All race/ethnicities and both genders will be included. Participants will be enrolled on a rolling basis from June 1, 2014-June 2, 2019. Participants will be involved in the study for approximately one year. The investigators anticipate a total of 1200 participants.
5. Subject Recruitment Methods and Privacy: Participants will be recruited through churches and other community settings. If eligible (see above), project staff will call potential participants within five days to verify eligibility and determine their interest in participating in the study.
6. Informed Consent Process: For those indicating an interest in participating, staff will visit potential participants at their home or a location of their choosing and administer the informed consent document. Study personnel for all phases of the project will provide a clear explanation of the project and invite questions. Our informed consent forms are written in a basic language. Interested participants will be asked to provide their signature on the informed consent forms. A copy of the signed consent will be provided for all participants. All forms will be read to participants to allay concerns about limited literacy. No non-English speaking or cognitively impaired participants will be recruited.
7. Research Procedures: The consort diagram (Figure 1) below provides an estimation and visual description of the recruitment and sampling frame.

   Fig 1: Consort diagram of enrollment
   1. Once informed consent documents are completed, participants (N=1200) will undergo the baseline assessment. Baseline, posttest, and exit assessments will consist of the same measures highlighted in Table 3.
   2. There will be three arms. For those randomized to the diabetes self management program (n=435), within two weeks of initial recruitment and baseline assessment, project staff will schedule the participant to attend a group Diabetes Self-management Program, a six week, lay lead and en evidence-based diabetes home self-management program (See Table 1, DSMP contents). Staff will arrange for the group sessions of the DSMP. One session will take place every other week. Upon completion of the DSMP program, approximately three month later, clinic navigation will be implemented. For those randomized to the Patient Navigation group, within two weeks of initial recruitment and baseline assessment, project staff will schedule the participant to meet with the Community Health Worker who will strategize about insuring that patients make their doctors' appointments as scheduled. The CHW/Patient Navigator will make at least 4 calls to each participant randomized to this group. For those randomized to the combined Community to Clinic Navigation, CCN (n=435), both of the activities for the Diabetes self management education group and the Patient navigation will be conducted. At month 5-6, the posttest will take place. To assess sustainability, 3-4 months later, navigation again will take place. An interviewer will complete the exit interview in month 10-11 using the same assessments. All throughout the intervention, standard medical visits will take place.

      Fig 2: Flow diagram of intervention and control activities by month

      Table 1: DSMP contents and conduct:

      Class Number Content/Objectives./Activities
      1. Diabetes: causes, diagnosis, incidence, and prevalence Discussion using a pancreas model and the handout "Understanding Diabetes". How to talk with your doctor and being a proactive patient. Goal setting
      2. Blood glucose testing, hyperglycemia, and hypoglycemia Discussion of the blood glucose-testing procedure, review of the handouts "Hyperglycemia" and "Hypoglycemia. Goal check in
      3. Eating right for diabetes, discussion of the food pyramid and dietary strategies ; Review of handouts. Goal check in
      4. Avoiding complications: Eye care, dental care, neuropathy, hypertension Discussion of appropriate eye care, dental care, kidney care. Review of how to talk with your doctor. Goal check in
      5. Getting active: review of physical activity and foot care. Goal check in
      6. Empowerment and goal check in. Class discussion.

      Table 2: Timeline

      Activity Q1 Q2 Q3 Q4 Staff training Recruitment, informed consent, enrollment, randomization Baseline medical record review/ interview 0 CCN arm participants receive DSM sessions (6 sessions total) and navigation to clinic X X Posttest 1 0 CCN arm Navigation X Exit interview 0 CCN= clinic to community navigation (intervention arm); DSM= diabetes self-management; X= intervention activity; 0= assessment
8. Resources: The research and intervention activities will be conducted in participants' homes, community sites, and the health clinics.
9. Potential Risks: The potential risks from participating in the study are very small. Some risk of pain from a finger prick or psychological upset could result from responding to interview questions or the emotional distress from questions about diabetes management. The most significant risk involves any threat to confidentiality. However, all project staff will be human subjects trained and have extensive experience maintaining participant confidentiality.
10. Safety Precautions: In each stage of the research, the investigators will make every effort to provide protection against risks. Study personnel will provide a clear explanation of the project and invite questions during enrollment. In the rare event that a participant experiences psychological distress resulting from the interview questions or from the intervention, our staff will contact Dr. Van Breeding, internal medicine physician at the MCHC. Dr. Breeding will consult with the participant, debrief and discuss the participant's concerns, and refer participants to any additional support. In addition, all project staff will receive training on how to respond to a participant who needs additional assistance with diabetes management.
11. Benefit vs. Risk Participation in the study involves little risk for subjects in comparison to the potential benefits of adopting improving diabetes outcomes. Participants in the intervention group will receive their usual care, plus navigation from a staff person at MCHC and an evidence-based diabetes self-management program at no cost. If they are not assigned to the intervention arm, they will receive their usual diabetes care. Given the disproportionate diabetes burden experienced by Appalachian populations, implementing and evaluating this novel, theory based intervention has the potential to save many lives while advancing intervention science.
12. Available Alternative Treatment(s): Participants will be randomized to the intervention (the standard of care plus navigation with a clinic employee and community-based navigation) OR will receive the standard treatment, which involves brief clinically-based consultation with the health care provider.
13. Research Materials, Records, and Privacy: Two sources of data will be collected: physiologic data collection (HbA1C levels, blood pressure, lipids, and BMI); and quantitative assessments (surveys). Table 3 highlights the specific data to be collected.

Table 3: Variables Data sources and collector Main outcomes HbA1C, blood pressure, lipids, waist circumference, BMI Additional outcomes: Self-management outcomes Medication taking, blood glucose testing, appointment adherence, diet, physical activity, foot and eye care.

Assessments by UK project staff Diabetes Empowerment Scale (self-efficacy), patient activation Assessments by UK project staff Sociodemographic, self-perceived health status, depression, Clinic attendance, assessments by UK project staff

14. Confidentiality Confidentiality of all data will be maintained by never linking paper or computer copy of data with the participants' names. A sheet with the participant's name, address, telephone number, and identification number will be kept by the Project Director and Principal Investigator separately in a locked file. Only staff members who are authorized to review files will be permitted access to the data. As part of our training, each lay health adviser and interviewer will be asked to sign a confidentiality pledge promising never to reveal, alter, or falsify survey data. This pledge is especially important in small, tight-knit rural communities. Data are held in password-protected computers and secure servers at University of Kentucky which have extensive firewalls and security measures. The investigator will keep all records (tapes, informed consent documents, and other records like completed questionnaires) for a minimum of six years after the completion of the study.

16. Costs to Subjects: N/A for program participation. Some costs associated with transportation may occur.

17. Data and Safety Monitoring: N/A 18. Subject Complaints: Participants will be asked to contact the investigator, Dr. Nancy Schoenberg at 859-323-8175 should they have any complaints. If they have any questions about their rights as a volunteer in this research, they will be asked to contact the staff in the Office of Research Integrity at the University of Kentucky at 859-257-9428 or toll free at 1-866-400-9428.

19. Research Involving Non-English Speaking Subjects or Subjects from a Foreign Culture: N/A 20. HIV/AIDS Research: N/A 20. PI-Sponsored FDA-Regulated Research: N/A

Two main revisions for this trial were implemented.

1. Timelines: Reduced the 18 month follow up to 9 months and then, ultimately, from 9 months to 6 months.
2. Data collection for several secondary outcomes:

   1. Data for HDL, LDL, cholesterol was not collected for two reasons:

1) lack of a scientific evidence base on the association between lipids and diabetes self-management and diabetes outcomes.

2) The extremely high cost of such data collection. b. We ceased collecting data on clinic attendance. At baseline, we collected data on clinic attendance within the standard guideline of 3 months. To our surprise, 87% of our sample had clinic appointments consistent with recommended guidelines. Thus, we could not realistically expect any significant improvements in subsequent time periods. Such a revelation, in conjunction with the cessation of clinical operations due to COVID, made clinic attendance data collection unnecessary and unfeasible. When the project began in 2017, the uninsured population of Appalachian Kentucky dropped from 25% to 6.7%. This coverage resulted in most participants adhering to the recommendations for clinic attendance.

Several significant events undermined the original data collection plan including:

* 24 month cessation of recruitment, data collection and intervention implementation due to COVID
* Episodic cessation of recruitment, data collection and intervention implementation due to COVID
* Major interruption of recruitment, data collection and intervention implementation due to natural disaster (flooding July 2022)
* Lack of NIH approval of two supplement requests to support data collection

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18+);
* Appalachian residence, no plans to relocate out of the area in the next 18 months,
* Willingness and ability to participate (i.e., no major cognitive impairment)
* HbA1c levels at least 6.5% or Diagnosis of Diabetes.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2018-04-29 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Schoenberg, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smalls BL, Adegboyega A, Combs E, Rutledge M, Westgate PM, Azam MT, De La Barra F, Williams LB, Schoenberg NE. The mediating/moderating role of cultural context factors on self-care practices among those living with diabetes in rural Appalachia. BMC Public Health. 2021 Oct 2;21(1):1784. doi: 10.1186/s12889-021-11777-7. PMID 34600524
- [Background] Smalls BL, Lacy ME, Adegboyega A, Hieronymus L, Bacha N, Nathoo T, Westgate PM, Azam T, Westneat S, Schoenberg NE. A New Look at Barriers to Clinical Care Among Appalachian Residents Living With Diabetes. Diabetes Spectr. 2023 Winter;36(1):14-22. doi: 10.2337/ds22-0001. Epub 2022 Nov 18. PMID 36818407
- [Background] Smalls BL, Azam T, Dunfee M, Westgate PM, Westneat SC, Schoenberg N. The relationship between psychosocial factors, self-care, and blood sugar in an Appalachian population. J Appalach Health. 2023 Jan 1;4(3):1-22. doi: 10.13023/jah.0403.01. eCollection 2023. PMID 38026048
- [Background] Smalls BL, Adegboyega A, Combs E, Travis EW, De La Barra F, Williams LB, Schoenberg N. Evaluating the Association Between Depressive Symptoms and Glycemic Control Among Residents of Rural Appalachia. J Appalach Health. 2023 Jan 1;4(3):39-55. doi: 10.13023/jah.0403.03. eCollection 2023. PMID 38026049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through churches and organizations in several KY counties in Appalachian Kentucky
Pre-assignment Details: 59 churches/organizations were randomized once they met the eligibility criteria. One church was never enrolled because it did not meet the eligibility criteria. Two churches/organizations dropped out mainly due to COVID issues.
Units Other Than Participants: Church/Organization
Groups:
- Diabetes Self-Management Program (DSMP) Only: Diabetes Self Management Program (DSMP) in a group setting: participants will attend a six week, evidence-based diabetes home self-management program. The goal of this arm of the project is to try to get participants to engage in better diabetes self-care (blood glucose testing, medication taking, diet, exercise, stress reduction, etc.).
  Participants will complete biometric data and surveys at 3, 6, and 9 months post randomization.
- Diabetes Self-Management Program (DSMP)Delayed: Groups randomized to DSMP Delayed will receive 6 weeks of DSMP classes after the 3 month post-test interview.
  Participants will complete biometric data and surveys at 3, 6, and 9 months post randomization.
- Tailored Patient Navigation (PN) Only: assisting patients in navigation to physician offices, allowing for standard of care to follow.
  trained Community Health Workers (CHW) will meet one-on-one with participants to assess the barriers experienced in adhering to medical appointments and will implement a navigation program accordingly.
  The goal of this arm of the project is to try to get participants to attend recommended medical appointments. PN has been shown to improve health behavior and increase self-efficacy, all with low costs.
Period: Overall Study
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP)Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Started | 198; 14 Church/Organization | 200; 15 Church/Organization | 120; 15 Church/Organization | 183; 15 Church/Organization
Completed | 150; 14 Church/Organization | 144; 13 Church/Organization | 91; 15 Church/Organization | 138; 15 Church/Organization
Not Completed | 48; 0 Church/Organization | 56; 2 Church/Organization | 29; 0 Church/Organization | 45; 0 Church/Organization
Not completed — Withdrawal by Subject | 36 | 29 | 11 | 27
Not completed — COVID | 0 | 23 | 0 | 0
Not completed — Participant moved from area | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 3 | 18 | 17
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Participant Removed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation | Total
Number analyzed (Participants) | 198 | 200 | 120 | 183 | 701
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (11.6) | 65.3 (9.3) | 61.9 (13.3) | 62.7 (11.2) | 63.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 121 | 76 | 116 | 449
  Male | 62 | 79 | 44 | 67 | 252
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 197 | 199 | 119 | 182 | 697
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 4 | 6
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 1 | 11 | 4 | 24
  White | 189 | 198 | 107 | 175 | 669
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 198 | 200 | 120 | 183 | 701

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c
Description: Changes in hemoglobin A1c (HbA1c) will be measured with a Bayer DCA 2000+ Analyzer (21), which has a test coefficient of variation < 5% consistent with requirements of the National Diabetes Data Group.
Time Frame: Baseline, month 3, month 6, month 9
Population: Number of observations for this particular outcome; i.e., contributed subject-level outcomes; Primary interest for DSMP and Delayed DSMP is baseline to 3 months, after 3 months, the Delayed DSMP group receives DSMP.
  For the PN and DSMP+PN study design, 9 month data were not collected
Measure: Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 198 | 200 | 120 | 183
percentage of glycated hemoglobin
  baseline to month 3: number analyzed (Participants) | 158 | 153 | 99 | 157
  baseline to month 3 | -0.37 (0.07) | -0.15 (0.08) | -0.31 (0.12) | -0.20 (0.10)
  baseline to month 6: number analyzed (Participants) | 158 | 149 | 93 | 139
  baseline to month 6 | -0.38 (0.08) | -0.37 (0.08) | -0.21 (0.14) | -0.20 (0.11)
  baseline to month 9: number analyzed (Participants) | 145 | 121 | 0 | 0
  baseline to month 9 | -0.40 (0.09) | -0.22 (0.10) |  |

2. Secondary Outcome: Change in Body Mass Index
Description: Change in calculated as a change in weight in kilograms divided by the square of height in meter.
Time Frame: Baseline, month 3, month 6, month 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg/m2
Groups:
- Tailored Patient Navigation (PN) Only: assisting patients in navigation to physician offices, allowing for standard of care to follow.
  Tailored Patient Navigation (PN) only: trained Community Health Workers (CHW) will meet one-on-one with participants to assess the barriers experienced in adhering to medical appointments and will implement a navigation program accordingly.
  The goal of this arm of the project is to try to get participants to attend recommended medical appointments. PN has been shown to improve health behavior and increase self-efficacy, all with low costs.
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 198 | 200 | 120 | 183
kg/m2
  baseline to month 3: number analyzed (Participants) | 158 | 153 | 99 | 157
  baseline to month 3 | -0.06 (0.10) | -0.23 (0.10) | -0.44 (0.13) | -0.14 (0.10)
  baseline to month 6: number analyzed (Participants) | 158 | 149 | 93 | 139
  baseline to month 6 | -0.05 (0.12) | -0.34 (0.13) | -0.57 (0.21) | -0.35 (0.17)
  baseline to month 9: number analyzed (Participants) | 144 | 121 | 0 | 0
  baseline to month 9 | -0.16 (0.14) | -0.41 (0.14) |  |

3. Secondary Outcome: Change in Waist Circumference
Description: Change in Waist circumference at the umbilical waist using the Tech-Med model cat. no. 4414.
Time Frame: Baseline, month 3, month 6, month 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: inches
Groups:
- Diabetes Self-Management Program (DSMP): Diabetes Self Management Program (DSMP) in a group setting: participants will attend a six week, evidence-based diabetes home self-management program. The goal of this arm of the project is to try to get participants to engage in better diabetes self-care (blood glucose testing, medication taking, diet, exercise, stress reduction, etc.).
  Participants will complete biometric data and surveys at 3, 6, and 9 months post randomization.
Arm/Group | Diabetes Self-Management Program (DSMP) | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 198 | 200 | 119 | 183
inches
  baseline to month 3: number analyzed (Participants) | 158 | 153 | 99 | 157
  baseline to month 3 | -0.25 (0.16) | -0.41 (0.16) | -0.54 (0.22) | -0.46 (0.18)
  baseline to month 6: number analyzed (Participants) | 155 | 149 | 93 | 139
  baseline to month 6 | -0.63 (0.18) | -0.89 (0.18) | -0.63 (0.29) | -0.99 (0.23)
  baseline to month 9: number analyzed (Participants) | 140 | 120 | 0 | 0
  baseline to month 9 | -1.09 (0.19) | -0.73 (0.19) |  |

4. Secondary Outcome: Number of Participants Attending a Clinic Visit
Description: Number of participants with a primary care provider that attended a clinic visit with that provider within the last 3 months.
Time Frame: Baseline
Population: Participants with a PCP that provided data for this outcome.
  Data only collected at baseline for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP)Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 128 | 140 | 83 | 98
Participants
  PCP Visit in last 3 months at baseline | 113 | 118 | 70 | 87
  No Visit to PCP in last 3 months at baseline | 15 | 22 | 13 | 11

5. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure will be reported as the average of two sphygmomanometer readings
Time Frame: Baseline, month 3, month 6, month 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 198 | 200 | 120 | 183
mm Hg
  baseline to month 3: number analyzed (Participants) | 158 | 153 | 99 | 157
  baseline to month 3 | -4.37 (1.56) | -0.47 (1.58) | -2.97 (1.95) | -3.86 (1.56)
  baseline to month 6: number analyzed (Participants) | 158 | 149 | 93 | 139
  baseline to month 6 | -4.22 (1.59) | 0.46 (1.63) | -6.60 (2.04) | -3.56 (1.66)
  baseline to month 9: number analyzed (Participants) | 145 | 121 | 0 | 0
  baseline to month 9 | -5.85 (1.75) | 1.02 (1.85) |  |

6. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure will be reported as the average of two sphygmomanometer readings
Time Frame: Baseline, month 3, month 6, month 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 198 | 200 | 120 | 183
mm Hg
  baseline to month 3: number analyzed (Participants) | 158 | 153 | 99 | 157
  baseline to month 3 | -2.25 (0.86) | -1.60 (0.87) | -3.01 (1.30) | -1.12 (1.04)
  baseline to month 6: number analyzed (Participants) | 158 | 149 | 93 | 139
  baseline to month 6 | -1.79 (0.87) | -1.69 (0.89) | -4.09 (1.33) | -1.07 (1.08)
  baseline to month 9: number analyzed (Participants) | 145 | 121 | 0 | 0
  baseline to month 9 | -2.95 (0.95) | -3.57 (1.01) |  |

7. Secondary Outcome: High Density Lipoprotein (HDL)
Description: blood will be drawn and HDL will be measured using a Cholestech LDX point of care machine. Data will be reported as the change in HDL over 18 months
Time Frame: Baseline to month 9
Population: Data not collected
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP)Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Low Density Lipoprotein (LDL)
Description: blood will be drawn and LDL will be measured using a Cholestech LDX point of care machine. Data will be reported as the change in LDL over 18 months
Time Frame: Baseline to month 9
Population: Data not collected
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP)Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Total Cholesterol
Description: blood will be drawn and Total cholesterol will be measured using a Cholestech LDX point of care machine. Data will be reported as the change in total cholesterol over 18 months
Time Frame: Baseline to month 9
Population: Data not collected
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP)Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Change in Physical Component Summary Score of SF-36
Description: The RAND SF-36 physical component summary (PCS) score is a domain summary score that is part of the 36-Item Short Form Health Survey (SF-36). Scores range from 0 - 100. Higher scores indicate better health or function. The PCS score is calculated by adding up standardized, weighted scores based on eight domains of health, including physical functioning and pain: Limitations in physical activities due to health problems, Bodily pain, and Vitality (energy and fatigue). Specific scoring details are provided in Taft et al. (2001).
Time Frame: Baseline, month 3, month 6, month 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Tailored Patient Navigation (PN) Only: assisting patients in navigation to physician offices, allowing for standard of care to follow.
  Tailored Patient Navigation (PN) only: Tailored Patient Navigation (PN) only: The goal of this arm of the project is to try to get participants to attend their recommended medical appointments. PN has been shown to improve health behavior and increase self-efficacy, all with low costs. We will have to add an additional eligibility criterion for this group-they have to be out of compliance with medical appointments. Most participants will need PN services, owing to missed, rescheduled, or infrequent appointments. This means not attending their office visits, as recommended, which typically is every 3 months. We will interact with them to verify attendance and, at times, to access patient medical records if needed.
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 197 | 199 | 120 | 182
score on a scale
  baseline to month 3: number analyzed (Participants) | 167 | 156 | 97 | 158
  baseline to month 3 | 0.29 (0.64) | -0.74 (0.67) | -1.39 (0.89) | 1.00 (0.70)
  baseline to month 6: number analyzed (Participants) | 159 | 150 | 93 | 140
  baseline to month 6 | 1.00 (0.69) | -0.40 (0.71) | 0.92 (0.93) | 1.05 (0.75)
  baseline to month 9: number analyzed (Participants) | 153 | 134 | 0 | 0
  baseline to month 9 | 0.28 (0.74) | -1.05 (0.79) |  |

11. Secondary Outcome: Change in Mental Component Summary Score of SF-36
Description: The RAND SF-36 mental component summary (MCS) score is a domain summary score that is part of the 36-Item Short Form Health Survey (SF-36). Scores range from 0 - 100. Higher scores indicating better mental health or function. The MCS score is calculated by adding up standardized, weighted scores based on eight domains of health, including physical functioning and pain: Limitations in physical activities due to health problems, Bodily pain, and Vitality (energy and fatigue). Specific scoring details are provided in Taft et al. (2001).
Time Frame: Baseline, month 3, month 6, month 9
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
Number analyzed (Participants) | 197 | 199 | 120 | 182
score on a scale
  baseline to month 3: number analyzed (Participants) | 167 | 156 | 97 | 158
  baseline to month 3 | 1.67 (0.74) | 1.73 (0.77) | 4.24 (1.03) | 1.21 (0.81)
  baseline to month 6: number analyzed (Participants) | 159 | 150 | 93 | 140
  baseline to month 6 | 1.56 (0.83) | 1.66 (0.85) | 4.05 (1.10) | 0.92 (0.89)
  baseline to month 9: number analyzed (Participants) | 153 | 134 | 0 | 0
  baseline to month 9 | 2.67 (0.84) | 1.82 (0.89) |  |

ADVERSE EVENTS:
Time Frame: 9 months
Description: Participant files were reviewed monthly from enrollment through the final follow up
Groups:
- DSMP AND Tailored Patient Navigation: Both group education classes and patient navigation
  DSMP AND Tailored Patient Navigation: DSMP AND Tailored Patient Navigation : Both group education classes and patient navigation
Arm/Group | Diabetes Self-Management Program (DSMP) Only | Diabetes Self-Management Program (DSMP) Delayed | Tailored Patient Navigation (PN) Only | DSMP AND Tailored Patient Navigation
All-Cause Mortality (participants affected / at risk) | 0/198 | 1/200 | 0/120 | 0/183
Serious Adverse Events (participants affected / at risk) | 0/198 | 0/200 | 0/120 | 0/183
Other Adverse Events (participants affected / at risk) | 0/198 | 0/200 | 0/120 | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03474731/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03474731/ICF_000.pdf